CLINICAL TRIAL: NCT04004273
Title: The Impact of Type 2 Diabetes and Exercise on Liver Fat Quality
Brief Title: Diabetes, Exercise and Liver Fat (DELIVER)
Acronym: (DELIVER)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: James King (Other)
Collaborators: University Hospitals, Leicester (Other); Nottingham University Hospitals NHS Trust (Other); University of Nottingham (Other)
Responsible Party: Sponsor-Investigator, James King, Chief Investigator, Loughborough University
Organization: Loughborough University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 241046
Record Dates: First submitted 2018-08-07; First posted 2019-07-02 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-10

CONDITIONS: Type 2 Diabetes Mellitus; Non-Alcoholic Fatty Liver Disease; Obesity; Insulin Resistance; Liver Diseases; Fatty Liver; Diabetes Mellitus; Glucose Metabolism Disorders; Glucose Intolerance; Metabolic Disease
Keywords: Type 2 diabetes; Non-alcohol fatty liver disease; Exercise; Saturated fat; MRI; Proton magnetic resonance spectroscopy
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Non-alcoholic Fatty Liver Disease; Obesity; Insulin Resistance; Liver Diseases; Fatty Liver; Diabetes Mellitus; Glucose Metabolism Disorders; Glucose Intolerance; Metabolic Diseases; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: A randomised control trial. Participants are randomised to an exercise group (treatment) or a control group (usual care/no treatment) for 6 weeks. Assessments occur at baseline and after 6 weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): Participants randomised to the exercise training intervention will complete 24 moderate-intensity exercise training sessions over the subsequent six weeks (four times per week; ~50 min per session). Each week, one exercise training session will be supervised by the research team, whilst three sessions will be unsupervised but monitored objectively using a heart rate monitor.
  Interventions: Behavioral: Exercise
- Control (No Intervention): Participants randomised to control will receive no interventions and will be requested to maintain their habitual lifestyle during the six week intervention phase

INTERVENTIONS:
Behavioral: Exercise — 24 moderate-intensity exercise training sessions over six weeks (four times per week; ~50 min per session)
  Arms: Exercise

SUMMARY:
This randomised controlled trial will determine if exercise (150 - 200 min per week, 6 weeks) can beneficially modify liver fat quality in non alcohol fatty liver disease patients with type 2 diabetes mellitus (n = 26, 13 per group). Liver fat quality will be assessed via magnetic resonance (3T) spectroscopy (1H-MRS) using validated methods.

DETAILED DESCRIPTION:
Verbal eligibility check

Prior to commencing the study, participants will be contacted via telephone and an initial verbal eligibility check will take place (approx. 30 min conversation). Following this, potentially eligible participants will be invited to visit the Sir Peter Mansfield Imaging Centre for study assessment visit one.

Assessment visit 1 - Sir Peter Mansfield Imaging Centre (University of Nottingham) Informed consent Before any study related procedures can take place, the participant must sign and date the most recent approved version of the Informed Consent Form. Before consent is obtained the responsible individual will ensure that the participant fully understands all aspects of the study. It will also be clearly stated that the participant is free to withdraw from the study at any time, for any reason, without prejudice to future care, and with no obligation to give the reason for withdrawal. If a participant withdraws from the study but does not withdraw their consent, then data already obtained may be used for the study. If a participant has withdrawn due to an adverse event, a medical professional will follow up as appropriate.

The consent form will be signed and dated based up on an informed decision. The consent process will be performed by someone who has received consent training, has been authorised by the Chief Investigator, and is named on the delegation of authority log. The original signed form will be retained at the study site and copy will be given to the participant. A third copy will be posted to the participant's GP.

Questionnaires

Participants will complete several pen and paper based questionnaires to assess their eligibility to participate in the study and to provide baseline study data. These will include the following:

* Physical Activity Readiness Questionnaire - to determine participants' readiness to exercise and/or contraindications
* Loughborough University Health Screen Questionnaire - to obtain an overview of participants' medical history, current medications and family history of disease
* Sir Peter Mansfield Imaging Centre Magnetic Resonance Safety Screening Form - to assess potential contraindications to MRI
* Demographics & contact details - to determine participants' date of birth, ethnicity and postal address
* Alcohol intake questionnaire - to determine participant's habitual alcohol intake in order to classify as non-alcoholic fatty liver disease.

Anthropometry, blood pressure and finger prick blood test Height, body mass and waist circumference will be measured using standard techniques and body mass index (BMI) will be calculated. Body fat percentage will be estimated using bioelectrical impedance analysis. Blood pressure will be assessed using an automated monitor after participants have sat quietly for 10 minutes (average of three measurements). A finger prick blood test will be taken to check preliminary eligibility (HbA1c) using a point-of-care device.

Magnetic resonance imaging (MRI) MRI data will be acquired using a 3T Philips Ingenia MRI scanner. Liver fat quality indices and total intrahepatocellular liver fat fractions will be determined using 1H-MRS via the quantification of individual lipid group peaks. Liver inflammation, visceral adipose tissue and subcutaneous abdominal adipose tissue will be measured via MRI. The techniques used to measure these outcomes have been validated and published previously.

Familiarisation with weighed food records and physical activity monitors Participants will be provided with a wrist worn (watch-like) physical activity monitor (GENEactiv) that they will wear 24 h/day for the next seven days. Participants will also be shown how to keep an accurate weighed food record and will be provided with food scales and diary to facilitate a three day record within the next seven days (two week and one weekend day).

After this session, MRI scans will be assessed to examine whether or not participants have an amount of liver fat that if high enough for inclusion in the study (> 5.56%). If liver fat is less than this then participants will not be permitted to participate. If liver fat is equal to or greater than this level then participants will be invited to attend study assessment visit two.

Assessment visit 2 - Leicester General Hospital (Leicester Diabetes Centre)

Fasting blood sample

Participants will be asked to attend the second study assessment visit having not eaten since the prior evening. These visits will therefore occur in the morning (before 10:30). At the start of this visit participants will provide a fasting venepuncture blood sample (40 mL blood) after having sat down for 10 minutes. This sample will be collected from an antecubital vein by an individual trained and experienced in phlebotomy. One blood bottle will be sent to hospital pathology labs for the analysis of glycated haemoglobin. The remaining samples will be spun immediately in a refrigerated centrifuge to obtain plasma/serum. These samples will subsequently be stored until the end of the trial within -80 degrees (celsius) freezers at the research sites. Following the last participants visit, samples will be transported to Loughborough University (at -80 degrees ) by a commercial courier. Samples will then be analysed in batch for:

* Lipids
* C-reactive protein
* Liver enzymes
* Glucose
* Insulin
* Nonesterifed fatty acids
* Hepatokines
* Inflammatory proteins

Medical evaluation and aerobic fitness A medical professional will take a full medical history from participants in order to identify any factors that may prohibit individuals from completing the study. A 12 lead ECG will also be performed. Finally, a symptom limited progressive treadmill exercise test will be undertaken on a treadmill. This test will require participants to exercise at increasingly harder intensities until volitional exhaustion. A clinical professional will monitor participants' blood pressure and ECG during this test which will be terminated if clinically indicated.

Randomisation After visit two participants will be randomised (1:1) to condition (exercise training or control). Randomisation will be performed by a trial statistician (see section 13 for additional details). The involvement of participants who are only completing Part A of the study will end at this point.

Six week intervention Participants randomised to control will receive no interventions during the six week intervention phase. During this time, control participants will be asked to not change any aspects of their lifestyles. Ahead of week five, participants will be posted a physical activity monitor to wear continuously during week five and six. Participants will also complete weighed food diaries during week five (two week days and one weekend day).

Participants randomised to exercise training will complete four exercise training sessions per week during the six week intervention. Each week, one session will be supervised by the research team whilst three sessions of brisk walking will be undertaken unsupervised by the participant. All exercise sessions will be composed of continuous moderate-intensity exercise and last 35 - 50 minutes in duration (depending on intervention week).

Assessment visit 3 (post-intervention) - Sir Peter Mansfield Imaging Centre (University of Nottingham) The assessments undertaken at visit three will be a repeat of those completed during visit one.

Assessment visit 4 (post-intervention) - Leicester General Hospital (Leicester Diabetes Centre) The assessments undertaken at visit four will be a repeat of those completed during visit two except that a medical examination will not be performed.

ELIGIBILITY:
Inclusion Criteria:

* Men
* ≥ 30 - ≤ 75 years of age
* Body mass index ≥ 27 - ≤ 45 kg/m2 (or ≥ 23 to 45 45 kg/m2 if south Asian)
* Waist circumference ≥ 94 cm (or ≥ 90 cm if south Asian)
* Clinically elevated liver fat (≥ 5.56% assessed via 1H-MRS)
* Participant is willing and able to give informed consent to participate
* Participant can communicate effectively in English
* Participant is able to meet the time demands of the study

Additional criteria for participants without T2DM:

• HbA1c > 6.0%

Additional criteria for participants with T2DM/prediabetes:

* Diagnosed T2DM or prediabetes
* Treatment via lifestyle or metformin only within the last 6 months
* HbA1c 6.0 - 10%
* Able to meet the time and physical demands encompassed within the exercise training intervention

Exclusion Criteria:

* Contraindications to magnetic resonance procedures
* Contraindications to exercise training
* Participating in regular purposeful exercise training of vigorous intensity - frequency greater than or equal to 3 sessions per week and intensity greater than or equal to 6.0 metabolic equivalents (METs)
* Weight instability or planned/ on-going dietary intervention
* Unable to communicate sufficiently in English
* Co-morbidity that the research team determine to be a contraindication to involvement
* Current smoker
* Uncontrolled hypertension - systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 100 mmHg

Additional criteria for participants with T2DM/prediabetes:

* Taking additional oral anti-diabetic medications to metformin e.g. SGLT2i, GLP-1RA, DPP4 inhibitors, TZDs within the last 6 months
* Taking insulin

Ages: 30 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2022-07-20 (Actual)

PRIMARY OUTCOMES:
Change in liver saturated lipid index (%) determined by proton magnetic resonance spectroscopy (1H-MRS) using a 3T MRI scanner | 2 measurements: Baseline, week 6
  Response to a six week exercise training intervention

SECONDARY OUTCOMES:
Change in Liver unsaturated lipid index (%) - measured using 1H-MRS | 2 measurements: Baseline, week 6
  Response to a six week exercise training intervention
Change in Liver polyunsaturated lipid index (%) - measured using 1H-MRS | 2 measurements: Baseline, week 6
  Response to a six week exercise training intervention
Change in total hepatic lipid composition (%) - measured using 1H-MRS | 2 measurements: Baseline, week 6
  Response to a six week exercise training intervention
Change in visceral adipose tissue - measured using magnetic resonance imaging (MRI) with a 3T Philips Ingenia MRI scanner | 2 measurements: Baseline, week 6
  Response to a six week exercise training intervention
Change in subcutaneous abdominal adipose tissue - measured using magnetic resonance imaging (MRI) with a 3T Philips Ingenia MRI scanner | 2 measurements: Baseline, week 6
  Response to a six week exercise training intervention
Change in body mass | 2 measurements: Baseline, week 6
  Body mass determined with scales. Response to a six week exercise training intervention
Change in body fat percentage | 2 measurements: Baseline, week 6
  Body fat percentage determined via bio-electrical impedance. Response to a six week exercise training intervention
Change in aerobic fitness (peak oxygen uptake) | 2 measurements: Baseline, week 6
  Treadmill based aerobic fitness test. Response to a six week exercise training intervention
Change in liver enzymes | 2 measurements: Baseline, week 6
  Response to a six week exercise training intervention. Measured in fasted venous plasma samples using enzymatic, colorimetric methods using a semi-automatic, bench-top analyser.
Change in glucose | 2 measurements: Baseline, week 6
  Response to a six week exercise training intervention. Measured in fasted venous plasma samples using enzymatic, colorimetric methods using a semi-automatic, bench-top analyser.
Change in insulin | 2 measurements: Baseline, week 6
  Response to a six week exercise training intervention. Measured in fasted venous plasma samples using a commercially available enzyme-linked immunosorbent assay (ELISA).
Change in lipids | 2 measurements: Baseline, week 6
  Response to a six week exercise training intervention. Measured in fasted venous plasma samples using enzymatic, colorimetric methods using a semi-automatic, bench-top analyser.
Change in HbA1c | 2 measurements: Baseline, week 6
  Response to a six week exercise training intervention. Measured in fasted venous plasma samples using enzymatic, colorimetric methods using a semi-automatic, bench-top analyser.
Change in homeostasis model assessment of insulin resistance (HOMA-IR; surrogate marker of hepatic insulin resistance) | 2 measurements: Baseline, week 6
  Response to a six week exercise training intervention. HOMA-IR will be calculated using fasted concentrations of plasma glucose and insulin.
Change in adipose tissue insulin resistance (ADIPO-IR; surrogate marker of adipose tissue insulin resistance) | 2 measurements: Baseline, week 6
  Response to a six week exercise training intervention. ADIPO-IR will be calculated using fasted concentrations of plasma insulin and non-esterified fatty acids.
Change in circulating Inflammatory proteins | 2 measurements: Baseline, week 6
  Response to a six week exercise training intervention. Measured in fasted venous plasma samples using a commercially available enzyme-linked immunosorbent assay (ELISA) and enzymatic, colorimetric methods using a semi-automatic, bench-top analyser.
Change in Hepatokines | 2 measurements: Baseline, week 6
  Response to a six week exercise training intervention. Measured in fasted venous plasma samples using a commercially available enzyme-linked immunosorbent assay (ELISA).
Change in objectively measured sedentary time - GENEactiv physical activity monitor | 2 measurements: Baseline, week 6
  monitor worn for 7 days on the wrist for 24 hrs
Change in objectively measured physical activity - GENEactiv physical activity monitor | 2 measurements: Baseline, week 6
  monitor worn for 7 days on the wrist for 24 hrs
Change in energy intake | 2 measurements: Baseline, week 6
  food diary - two weekdays and one weekend day. Response to a six week exercise training intervention
Change in macronutrient intake | 2 measurements: Baseline, week 6
  food diary - two weekdays and one weekend day. Response to a six week exercise training intervention

CONTACTS AND LOCATIONS:
Overall Officials: James A King, PhD, Principal Investigator — Loughborough University; Guruprasad P Aithal, PhD, Principal Investigator — Nottingham Biomedical Research Centre; David Webb, PhD, Principal Investigator — Leicester Diabetes Research Centre; Penny Gowland, PhD, Principal Investigator — Sir Peter Mansfield Imaging Centre
Locations (4):
- United Kingdom (4):
  - University Hospitals of Leicester Nhs Trust, Leicester, East Midlands
  - NIHR Clinical Research Network, Leicester, East Midlands
  - Sir Peter Mansfield Imaging Centre, Nottingham, East Midlands
  - Nottingham University Hospitals Nhs Trust, Nottingham, East Midlands

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2021-09-23): https://cdn.clinicaltrials.gov/large-docs/73/NCT04004273/Prot_002.pdf
  • Statistical Analysis Plan (2018-08-06): https://cdn.clinicaltrials.gov/large-docs/73/NCT04004273/SAP_001.pdf